CLINICAL TRIAL: NCT06885749
Title: Clinical and Psychosocial Characteristics of Adolescent Patients With Non-Suicidal Self-Injury
Status: Enrolling by invitation | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20232397-F-1
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-05

CONDITIONS: Non-suicidal Self-injury (NSSI); Adolescent; Depression
Keywords: Non-Suicidal Self-Injury; Adolescent; Depression; Psychosocial Characteristics
MeSH Terms: conditions — Self-Injurious Behavior; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case Study Group: Outpatients or inpatients who meet the ICD-11 criteria for emotional and behavioral disorders typically originating in childhood and adolescence; aged 12-18 years; exhibiting non-suicidal self-injury behaviors
- Case Control Group: Outpatients or inpatients who meet the ICD-11 criteria for emotional and behavioral disorders typically originating in childhood and adolescence; aged 12-18 years; no non-suicidal self-injury behaviors
- Healthy Control Group: Healthy adolescents

SUMMARY:
The overall objective of this study is to explore the social and clinical psychological characteristics of adolescents with depression accompanied or not accompanied by non-suicidal self-harm.

This is an observational study. A total of 90 cases were included, with 30 cases in each of the case study group, case control group and healthy control group.

DETAILED DESCRIPTION:
This project aims to explore the socio-psychological characteristics of children and adolescents with emotional disorders, with or without non-suicidal self-injury (NSSI). The study is designed as an observational research, enrolling a total of 90 cases divided into three groups: the case study group, the case control group, and the healthy control group, with 30 cases in each group.

The inclusion criteria for the case study group are: outpatients or inpatients who meet the ICD-10 criteria for emotional and behavioral disorders typically originating in childhood and adolescence; aged 12-18 years; exhibiting non-suicidal self-injury behaviors; and having obtained informed consent from the patients or their guardians, with signed informed consent forms. The inclusion criteria for the case control group are similar to those of the case study group, but require no history of non-suicidal self-injury. The inclusion criteria for the healthy group are: not meeting any ICD-10 diagnostic criteria for mental disorders; aged 12-18 years; no history of non-suicidal self-injury; and informed consent obtained from both the participants and their guardians.

Exclusion criteria include: currently having severe physical illnesses that researchers deem unsuitable for participation in this study; meeting ICD-10 Axis I diagnostic criteria for other mental disorders; having a history of suicidal behavior; and other conditions judged by researchers as unsuitable for participation in the study.

Outcome assessment is conducted through observational clinical research. After enrollment, participants undergo multiple questionnaire assessments, including the Hamilton Depression Scale, Hamilton Anxiety Scale, Adolescent Non-Suicidal Self-Injury and Function Scale (ANSAQ), Prosocial Tendency Measure for Adolescents (PTM), Center for Epidemiological Studies Depression Scale for Children (CES-DC), Self-Rating Anxiety Scale (SAS), Self-Rating Scale of Systemic Family Dynamics (SSFD), Chinese Big Five Personality Inventory Brief Version (CBF-PI-15), Perceived Social Support Scale (PSSS), Hong Kong Psychological Resilience Scale for Adolescents (HKRA), and Self-Compassion Scale (SCS). The primary outcome measure is the difference in scores on the Prosocial Tendency Measure for Adolescents among the case study group, case control group, and healthy control group. Secondary outcome measures include differences in scores on the aforementioned other questionnaires among the three groups.

Statistical analysis is performed using SPSS 23.0 statistical software. All statistical tests are two-sided, with a P-value of less than or equal to 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* meet the ICD-11 criteria for emotional and behavioral disorders typically originating in childhood and adolescence; aged 12-18 years; exhibiting non-suicidal self-injury behaviors; having obtained informed consent from the patients or their guardians, with signed informed consent forms.

Exclusion Criteria:

* currently having severe physical illnesses that researchers deem unsuitable for participation in this study; meeting ICD-11 Axis I diagnostic criteria for other mental disorders; and other conditions judged by researchers as unsuitable for participation in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Outpatients or inpatients at Xijing Hospital, the First Affiliated Hospital of the Air Force Medical University, Xi'an, China.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the differences in score on the Prosocial Tendency Measure for Adolescents among the case study group, case control group, and healthy control group. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Xijing Hospital, Xi'an, Shaanxi, China